CLINICAL TRIAL: NCT05238610
Title: Prospective Registry of Elderly Patients With ESUS to Evaluate the Role of Covert Atrial Fibrillation and Patent Foramen Ovale
Brief Title: Prospective Registry of Elderly ESUS With PFO
Acronym: COACH_ESUS
Status: Recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: National Evidence-Based Healthcare Collaborating Agency (Other Government)
Responsible Party: Principal Investigator, Sun U. Kwon, Professor, Asan Medical Center
Other Study IDs: COACH_ELDERLY_ESUS_NECA_2021
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Embolic Stroke of Undetermined Source
Keywords: insertable loop recorder; patent foramen ovale; patent foramen ovale closure; elderly
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: intervention group: This group will receive PFO-closure and standard antiplatelet treatment PFO-closure will be performed after 3-6 months of observation and monitoring for paroxysmal atrial fibrillation Standard antiplatelet treatment will be prescribed - aspirin 100mg and clopidogrel 75mg, once daily, principally. However, the final decision of antiplatelet treatment will be made by the physician. If paroxysmal atrial fibrillation is detected, anticoagulation will be considered.
  Intervention : PFO closure Drug: aspirin 100mg/day Drug: clopidogrel 75mg/day
  Interventions: Procedure: PFO closure
- Active comparator: control group: This group will receive standard antiplatelet treatment only Dual antiplatelet treatment with Aspirin 100mg and Clopidogrel 75mg, once daily, or single antiplatelet treatment with those agents can be considered. If paroxysmal atrial fibrillation is detected, anticoagulation will be considered.
  Drug: aspirin 100mg/day Drug: clopidogrel 75mg/day

INTERVENTIONS:
Procedure: PFO closure — PFO-closure will be performed after 3-6 month of observation and monitoring for paroxysmal atrial fibrillation
  Groups: Experimental: intervention group

SUMMARY:
Patent foramen ovale (PFO) is associated with an increased risk of stroke. PFO-closure was effective in preventing stroke in young stroke patients less than age 60 presented as an embolic stroke of undetermined source (ESUS). However, the benefit of PFO-closure in elderly ESUS patients is not clear. The investigators designed this prospective register-based observational study to verify the efficacy of PFO-closure in elderly ESUS patients with high-risk PFO, older than 60 years

DETAILED DESCRIPTION:
The COACH-ELDERLY ESUS study is a multicenter, prospective, registry-based, observational study in elderly ESUS patients with high-risk PFO treated with PFO-closure + standard antiplatelet treatment or standard antiplatelet treatment only in 20 centers in Korea.

Patients will receive an insertable loop recorder (ILR) to monitor paroxysmal atrial fibrillation. In cases, which are unavailable for ILR, recurrent EKG or Holter monitoring will be done based on the clinician's decision. Based on the attending physicians' decision with a multi-disciplinary approach, patients will receive PFO-closure with standard antiplatelet treatment or standard antiplatelet treatment only.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 60 years-old
2. Patients diagnosed as ESUS within 180 days from onset
3. PFO found from TTE or TEE, which attributed to the ischemic stroke
4. Patients or their legal representative agreed to participate

Exclusion Criteria:

1. Patients with transient ischemic attack
2. Patients with ischemic stroke at the vascular territory with significant stenosis
3. Patients with high risk cardioembolic stroke detected from EKG, Holter monitoring or echocardiography
4. Patients with other causes which may cause stroke (i.e. vasculitis, dissection, vasospasm, drug related or Moyamoya disease)
5. Patients with active cancer
6. Patients who need long term anticoagulation
7. Patients who have side effect on antiplatelet treatment
8. Patients with active internal bleeding
9. Patients who refuse to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly ESUS patients
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
ischemic stroke recurrence | at least 1 year
  Time to occurrence of ischemic stroke after registration

SECONDARY OUTCOMES:
MACE | at least 1 year
  Time to major cardiovascular event after registration
Hemorrhagic stroke | at least 1 year
  Time to hemorrhagic stroke after registration
Vascular death | at least 1 year
  Time to vascular death after registration
Myocardial infarction | at least 1 year
  Time to myocardial infarction
Atrial fibrillation after registration | at least 1 year
  Time to atrial fibrillation after registration
Atrial fibrillation lasting more than 2 or 6 min after registration | at least 1 year
  Time to atrial fibrillation lasting more than 2 or 6 min after registration
Major bleeding | at least 1 year
  Time to major bleeding event after registration

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kwon H, Lee PH, Song JK, Kwon SU, Kang DW, Kim JS. Patent Foramen Ovale Closure in Old Stroke Patients: A Subgroup Analysis of the DEFENSE-PFO Trial. J Stroke. 2021 May;23(2):289-292. doi: 10.5853/jos.2021.00647. Epub 2021 May 31. No abstract available. PMID 34102766
- [Background] Park S, Oh JK, Song JK, Kwon B, Kim BJ, Kim JS, Kang DW, Chang JY, Lee JS, Kwon SU. Transcranial Doppler as a Screening Tool for High-Risk Patent Foramen Ovale in Cryptogenic Stroke. J Neuroimaging. 2021 Jan;31(1):165-170. doi: 10.1111/jon.12783. Epub 2020 Sep 8. PMID 32896963
- [Background] Lee PH, Song JK, Kim JS, Heo R, Lee S, Kim DH, Song JM, Kang DH, Kwon SU, Kang DW, Lee D, Kwon HS, Yun SC, Sun BJ, Park JH, Lee JH, Jeong HS, Song HJ, Kim J, Park SJ. Cryptogenic Stroke and High-Risk Patent Foramen Ovale: The DEFENSE-PFO Trial. J Am Coll Cardiol. 2018 May 22;71(20):2335-2342. doi: 10.1016/j.jacc.2018.02.046. Epub 2018 Mar 12. PMID 29544871
- [Background] Kim BJ, Kim NY, Kang DW, Kim JS, Kwon SU. Provoked right-to-left shunt in patent foramen ovale associates with ischemic stroke in posterior circulation. Stroke. 2014 Dec;45(12):3707-10. doi: 10.1161/STROKEAHA.114.007453. Epub 2014 Oct 30. PMID 25358696
- [Background] Kim BJ, Sohn H, Sun BJ, Song JK, Kang DW, Kim JS, Kwon SU. Imaging characteristics of ischemic strokes related to patent foramen ovale. Stroke. 2013 Dec;44(12):3350-6. doi: 10.1161/STROKEAHA.113.002459. Epub 2013 Sep 26. PMID 24072002
- [Background] Jung JM, Lee JY, Kim HJ, Do Y, Kwon SU, Kim JS, Song JK, Kang DW. Patent foramen ovale and infarct volume in cryptogenic stroke. J Stroke Cerebrovasc Dis. 2013 Nov;22(8):1399-404. doi: 10.1016/j.jstrokecerebrovasdis.2013.04.034. Epub 2013 Jun 5. PMID 23747019
- [Background] Lee JY, Song JK, Song JM, Kang DH, Yun SC, Kang DW, Kwon SU, Kim JS. Association between anatomic features of atrial septal abnormalities obtained by omni-plane transesophageal echocardiography and stroke recurrence in cryptogenic stroke patients with patent foramen ovale. Am J Cardiol. 2010 Jul 1;106(1):129-34. doi: 10.1016/j.amjcard.2010.02.025. Epub 2010 May 13. PMID 20609660